CLINICAL TRIAL: NCT06014619
Title: Clinical Presentation and Surgical Outcomes in Patients With Skin Disorders Treated With Mohs Micrographic Surgery and Slow Mohs.
Brief Title: Complications and Recurrences After Mohs Micrographic Surgery and Slow Mohs
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0043
Record Dates: First submitted 2023-08-15; First posted 2023-08-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Skin Cancer; Complication; Complication of Surgical Procedure; Complication,Postoperative; Recurrence; Recurrent Disease; Cutaneous Squamous Cell Carcinoma; Basal Cell Carcinoma; Lentigo Maligna; Lentigo Maligna Melanoma
Keywords: Clinical presentation; Outcomes; Mohs micrographic surgery; Slow Mohs; Micrographic surgery
MeSH Terms: conditions — Skin Neoplasms; Postoperative Complications; Recurrence; Carcinoma, Basal Cell; Hutchinson's Melanotic Freckle | interventions — Mohs Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mohs Micrographic Surgery: Patients treated with Mohs Micrographic Surgery in the dermatology department of Maastricht University Medical Center +, Maastricht, the Netherlands
  Interventions: Procedure: Mohs surgery
- Slow Mohs: Patients treated with Slow Mohs in the dermatology department of Maastricht University Medical Center +, Maastricht, the Netherlands
  Interventions: Procedure: Slow Mohs surgery

INTERVENTIONS:
Procedure: Mohs surgery — Treatment of a skin disease by Mohs micrographic surgery technique (frozen sections).
  Other Names: Mohs micrographic surgery; MMS; Mohs
  Groups: Mohs Micrographic Surgery
Procedure: Slow Mohs surgery — Treatment of a skin disease by Slow Mohs technique (formalin fixation and paraffin-embedded sections).
  Other Names: Slow Mohs
  Groups: Slow Mohs

SUMMARY:
Mohs micro-graphic surgery (Mohs) is a tissue-sparing, surgical treatment for different types of skin cancer (e.g. basal cell carcinoma, squamous cell carcinoma, lentigo maligna (melanoma). It is a procedure performed with frozen sections. Slow Mohs, a variant of micro-graphic surgery, is performed by formalin fixation and paraffin-embedded sections. Both in Mohs and Slow Mohs tumor margins are assessed to achieve complete removal. This study aims to investigate the clinical presentation and outcomes (i.e. complications and recurrence rates) in patients treated with Mohs or Slow Mohs in the dermatology department of the Maastricht University Medical Center+ in Maastricht, the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* patients with a cutaneous lesion with an indication for Mohs micrographic surgery or Slow Mohs
* patients who received a treatment with either Mohs or Slow Mohs between 1 july 2017 and 1 july 2023 at the dermatology department of the Maastricht University Medical Center+.

Exclusion Criteria:

* None.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications | Within 1 month after completion of the surgical intervention.
  The incidence of complications after Mohs and Slow Mohs, expressed as absolute numbers and percentages.
Incidence of recurrence | Up to 5 year after completion of the surgical intervention.
  The incidence of complications after Mohs and Slow Mohs, expressed as absolute numbers and percentages. Recurrence is defined as disease relapse after completion of treatment.

SECONDARY OUTCOMES:
Hazard ratio of predisposing factors for complications | Within 1 month after completion of the surgical intervention.
  Predisposing factors (patient- and tumor characteristics) for complications after Mohs and Slow Mohs, expressed in Hazard Ratio's and 95% confidence intervals. It is not possible to define the predisposing factors in advance, because this is currently unknown. We hypothesize the presence of diabetes, tobacco use and medication use to be predisposing factors for complications.
Hazard ratio of predisposing factors for recurrence | Up to 5 year after completion of the surgical intervention.
  Predisposing factors (patient- and tumor characteristics) for recurrences after Mohs and Slow Mohs, expressed in Hazard Ratio's and 95% confidence intervals. It is not possible to define the predisposing factors in advance, because this is currently unknown. We hypothesize incomplete treatment, worse prognostic tumor factors (Stage III of IV, presence of perineural invasion or lymphovascular invasion) to be predisposing factors for recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: K Mosterd, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Lee CB, Roorda BM, Wakkee M, Voorham Q, Mooyaart AL, de Vijlder HC, Nijsten T, van den Bos RR. Recurrence rates of cutaneous squamous cell carcinoma of the head and neck after Mohs micrographic surgery vs. standard excision: a retrospective cohort study. Br J Dermatol. 2019 Aug;181(2):338-343. doi: 10.1111/bjd.17188. Epub 2018 Oct 28. PMID 30199574
- [Background] Lacerda PN, Lange EP, Luna NM, Miot HA, Nogueira VSN, Abbade LPF. Recurrence rate of basal cell carcinoma among different micrographic surgery techniques: systematic review with meta-analysis. J Eur Acad Dermatol Venereol. 2022 Aug;36(8):1178-1190. doi: 10.1111/jdv.18048. Epub 2022 Apr 1. PMID 35274381
- [Background] Cook JL, Perone JB. A prospective evaluation of the incidence of complications associated with Mohs micrographic surgery. Arch Dermatol. 2003 Feb;139(2):143-52. doi: 10.1001/archderm.139.2.143. PMID 12588220
- [Background] Nemer KM, Ko JJ, Hurst EA. Complications After Mohs Micrographic Surgery in Patients Aged 85 and Older. Dermatol Surg. 2021 Feb 1;47(2):189-193. doi: 10.1097/DSS.0000000000002452. PMID 32796326
- [Background] Merritt BG, Lee NY, Brodland DG, Zitelli JA, Cook J. The safety of Mohs surgery: a prospective multicenter cohort study. J Am Acad Dermatol. 2012 Dec;67(6):1302-9. doi: 10.1016/j.jaad.2012.05.041. Epub 2012 Aug 11. PMID 22892283
- [Background] Alam M, Ibrahim O, Nodzenski M, Strasswimmer JM, Jiang SI, Cohen JL, Albano BJ, Batra P, Behshad R, Benedetto AV, Chan CS, Chilukuri S, Crocker C, Crystal HW, Dhir A, Faulconer VA, Goldberg LH, Goodman C, Greenbaum SS, Hale EK, Hanke CW, Hruza GJ, Jacobson L, Jones J, Kimyai-Asadi A, Kouba D, Lahti J, Macias K, Miller SJ, Monk E, Nguyen TH, Oganesyan G, Pennie M, Pontius K, Posten W, Reichel JL, Rohrer TE, Rooney JA, Tran HT, Poon E, Bolotin D, Dubina M, Pace N, Kim N, Disphanurat W, Kathawalla U, Kakar R, West DP, Veledar E, Yoo S. Adverse events associated with mohs micrographic surgery: multicenter prospective cohort study of 20,821 cases at 23 centers. JAMA Dermatol. 2013 Dec;149(12):1378-85. doi: 10.1001/jamadermatol.2013.6255. PMID 24080866
- [Background] Basu P, Goldenberg A, Cowan N, Eilers R, Hau J, Jiang SIB. A 4-year retrospective assessment of postoperative complications in immunosuppressed patients following Mohs micrographic surgery. J Am Acad Dermatol. 2019 Jun;80(6):1594-1601. doi: 10.1016/j.jaad.2018.11.032. Epub 2018 Nov 28. PMID 30502411
- [Background] Patel SA, Liu JJ, Murakami CS, Berg D, Akkina SR, Bhrany AD. Complication Rates in Delayed Reconstruction of the Head and Neck After Mohs Micrographic Surgery. JAMA Facial Plast Surg. 2016 Sep 1;18(5):340-6. doi: 10.1001/jamafacial.2016.0363. PMID 27227423
- [Background] Huether MJ, Griego RD, Brodland DG, Zitelli JA. Clindamycin for intraincisional antibiotic prophylaxis in dermatologic surgery. Arch Dermatol. 2002 Sep;138(9):1145-8. doi: 10.1001/archderm.138.9.1145. PMID 12224974
- [Background] Rogers HD, Desciak EB, Marcus RP, Wang S, MacKay-Wiggan J, Eliezri YD. Prospective study of wound infections in Mohs micrographic surgery using clean surgical technique in the absence of prophylactic antibiotics. J Am Acad Dermatol. 2010 Nov;63(5):842-51. doi: 10.1016/j.jaad.2010.07.029. Epub 2010 Aug 30. PMID 20800320
- [Background] Maragh SL, Brown MD. Prospective evaluation of surgical site infection rate among patients with Mohs micrographic surgery without the use of prophylactic antibiotics. J Am Acad Dermatol. 2008 Aug;59(2):275-8. doi: 10.1016/j.jaad.2008.03.042. PMID 18638628
- [Background] Xia Y, Cho S, Greenway HT, Zelac DE, Kelley B. Infection rates of wound repairs during Mohs micrographic surgery using sterile versus nonsterile gloves: a prospective randomized pilot study. Dermatol Surg. 2011 May;37(5):651-6. doi: 10.1111/j.1524-4725.2011.01949.x. Epub 2011 Apr 1. PMID 21457390